CLINICAL TRIAL: NCT01891045
Title: Addiction Treatment Dropout Prevention - Impact of Online Patient Feedback (OQ-45.2) to Therapist
Brief Title: Impact of Online Patient Feedback (OQ) to Therapist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Espen Walderhaug, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OQ45-11-1
Record Dates: First submitted 2012-07-06; First posted 2013-07-02 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Drug Addiction; Drug Abuse
Keywords: Psychotherapy; Drug addiction; Drop-out; OQ-45.2; Clinical trial; Randomized Controlled Trail
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Patients merely monitored on background variables to function as a baseline of comparison
- Prediction (Active Comparator): Patients randomized to this condition completes the OQ-45.2 weekly, but the reports are withheld from therapists and patients.
  Interventions: Behavioral: OQ-45.2 no feedback
- Intervention (Experimental): Patients and therapists uses the feedback-system as intended, with real-time feedback to the therapist and full use of the suggested interventions
  Interventions: Behavioral: OQ-45.2

INTERVENTIONS:
Behavioral: OQ-45.2 no feedback — Completion of the OQ-45.2 before each session, but no feedback to therapists or patients
  Arms: Prediction
Behavioral: OQ-45.2 — Completion of the OQ-45.2 with real-time feedback to the therapist and full use of the suggested interventions every week of the treatment program
  Arms: Intervention

SUMMARY:
Dropout represents one of the largest problems in substance abuse treatment. International and Nordic research show that only 20 - 40 % of substance abusers complete treatment as intended. At the same time, one of the most consistent factors of favourable post-treatment outcome is treatment completion. In spite of the serious and continuous challenge dropout represents the phenomena is not well understood and there is a need to explore more of the factors that influence dropout and how it can be counteracted. As also stated: "…effective methods for reducing the problem of dropouts from treatment is one more area in need of further research" (NOU 2003:4, s 77).

For the general field of mental health one of the most important innovations involves providing therapists with patient feedback about their progress. The most well-established and widely researched feedback system is the Outcome Questionnaire (OQ-45.2). The system has been shown to improve treatment outcomes, including reduced treatment dropout and length of treatment, but the system is yet to be utilized with a substance abusing patient group. The aim of the present study is to examine the usefulness of OQ-45.2 with substance abusing patients.

DETAILED DESCRIPTION:
Hypotheses and research questions

1. The OQ-45.2 feedback will be effective in identifying patients at risk of dropout of substance abuse treatment.

1a. The condition were feedback is withheld from the therapist, will correctly identify patients who will dropout.

Research Question: Is there variation in the accuracy of dropout prediction as a function of age, gender differences or type of substance abuse?

2. The OQ-45.2 feedback will be effective in reducing dropout in outpatient substance abuse treatment.

2a. The feedback condition will result in less dropout than the no-feedback condition.

Research Question: Is there a variation in the OQ-45.2 preventive dropout effect due to age, gender or type of substance abuse?

3. The OQ-45.2 feedback will shorten length of inpatient substance abuse treatment.

3a. The feedback condition will identify patients who are ready to terminate therapy.

Research Question: Is there variation in identification of patients ready to terminate as a function of age, gender differences or type of substance abuse?

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of addiction, F10-19, using the International Classification of Diseases, admitted in 2011-2014 for treatment at the department of addiction treatment - youth, Oslo University Hospital

Exclusion Criteria:

* Ongoing psychoses, severe language difficulties

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2011-07-01; Primary Completion 2014-11-01 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Drop-out from residential SUD treatment | Four years
  Exit reason from residential Substance Use Disorder treatment (Drop-out or completed as planned)

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Department of addiction treatment- youth, Oslo
  - Oslo University Hospital - Department of addiction treatment youth, Oslo

REFERENCES:
- [Result] Amble I, Gude T, Stubdal S, Oktedalen T, Skjorten AM, Andersen BJ, Solbakken OA, Brorson HH, Arnevik E, Lambert MJ, Wampold BE. Psychometric properties of the outcome questionnaire-45.2: the Norwegian version in an international context. Psychother Res. 2014;24(4):504-13. doi: 10.1080/10503307.2013.849016. Epub 2013 Nov 5. PMID 24188797
- [Result] Brorson HH, Arnevik EA, Rand K. Predicting Dropout from Inpatient Substance Use Disorder Treatment: A Prospective Validation Study of the OQ-Analyst. Subst Abuse. 2019 Aug 15;13:1178221819866181. doi: 10.1177/1178221819866181. eCollection 2019. PMID 31452601